CLINICAL TRIAL: NCT03668015
Title: Xylitol and Sorbitol Effects on the Microbiome of Saliva and Plaque
Brief Title: Xylitol and Sorbitol Effects on the Oral Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Collaborators: J. Craig Venter Institute (Other)
Responsible Party: Principal Investigator, Reisha Rafeek, Senior Lecturer, The University of The West Indies
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CRP.3.MAR14.7
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Human Microbiome
Keywords: caries; bacteria; saliva; plaque; microbial ecology
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Xylitol then sorbitol gum) (Experimental): Subjects were randomly allocated to a group and entered a 4-week "washout period" during which no gum was chewed, followed by a 3-week treatment period (treatment period 1) during which Group A used Xylitol gum.(2 gum pieces, 3 times daily after meals for 6 minutes).Then underwent another 4-week washout period before entering treatment period 2 during which Group A used Gum Sorbitol
  Interventions: Other: Xylitol then Sorbitol gum
- Group B (Sorbitol then xylitol gum) (Experimental): Subjects were randomly allocated to a group and entered a 4-week "washout period" during which no gum was chewed, followed by a 3-week treatment period (treatment period 1) during which Group B used sorbitol gum. Group B used Gum Sorbitol (2 gum pieces, 3 times daily after meals for 6 minutes).Then underwent another 4-week washout period before entering treatment period 2 during which Group B used Gum xylitol
  Interventions: Other: Sorbitol then Xylitol gum

INTERVENTIONS:
Other: Xylitol then Sorbitol gum — Xylitol gum contains 70% xylitol in addition to gum base, natural flavors, soy lecithin, gum arabic, titanium dioxide, carnuba wax. Sorbitol gum was similar except that xylitol was replaced by 63% sorbitol and 2% maltitol and aspartame was included.
  Arms: Group A (Xylitol then sorbitol gum)
Other: Sorbitol then Xylitol gum — Sorbitol gum was similar except that xylitol was replaced by 63% sorbitol and 2% maltitol and aspartame was included. Xylitol gum contains 70% xylitol in addition to gum base, natural flavors, soy lecithin, gum arabic, titanium dioxide, carnuba wax.
  Arms: Group B (Sorbitol then xylitol gum)

SUMMARY:
Chewing gum containing xylitol may help prevent caries by reducing levels of mutans streptococci (MS) and lactobacilli in saliva and plaque. Very little is known about other species which are possibly beneficial to oral health. In this study, the investigators employed high-throughput sequencing of the 16S ribosomal ribonucleic acid (rRNA) gene to profile microbial communities of saliva and plaque following short-term consumption of xylitol and sorbitol containing chewing gum. Participants (n = 30) underwent a washout period and were randomly assigned to one of two groups. Each group chewed either xylitol or sorbitol gum for 3 weeks, before undergoing a second four-week washout period after which they switched to the alternate gum for three weeks.

DETAILED DESCRIPTION:
Subjects: Study protocols were approved by the Ethics Committees of the UWI, St. Augustine. Thirty healthy volunteers from The University of the West Indies (UWI), St. Augustine, Trinidad were enrolled in the study. To be eligible, subjects must have had at least 20 teeth, provided written informed consent and been willing to comply with study procedures. Subjects with systemic, infectious or inflammatory diseases or taking medicines, antibiotics or fluoride in the last month, habitual consumers of xylitol / sorbitol-containing products and mouth rinses, with abnormal salivary flow (<1ml / min), pregnant, on contraceptive pills, or with abnormal dietary habits were excluded. Consent obtained at the initial visit was verified at the second visit, prior to sample collection. The subjects were examined in the dental chair after thorough medical and dental histories were recorded. The clinical examination involved examination of the soft tissues and then dental hard tissue charting for presence of decayed, missing or filled teeth. No radiographs were used. The presence of untreated dental caries or periodontitis were not used as exclusion criteria. The decayed, missing, and filled teeth for each individual at the initial visit was documented for calculation of the index of decayed-missing-filled permanent teeth (DMFT) score.

Chewing gums: Xylitol gum (Epic Spearmint; 1.5g/pellet) designated Gum X contains 70% xylitol in addition to gum base, natural flavors, soy lecithin, gum arabic, titanium dioxide, carnuba wax. Gum S (Eclipse Spearmint), was similar except that xylitol was replaced by 63% sorbitol and 2% maltitol and aspartame was included. Gums were packed in colour-coded containers. Codes were kept confidential from the participants and researchers who interacted with them until study completion.

Study design: This prospective cross-over, double-blind, randomised study lasted 14 weeks (March - June, 2015). Throughout, subjects were instructed not to use mouthwashes or xylitol products, to consume a normal diet, continue their usual tooth brushing and to report use of antimicrobial medications. Subjects reporting the latter were dropped.

Subjects were randomly allocated to two groups, A and B (see Figure 1). Both groups entered a 4-week "washout period" during which no gum was chewed, followed by a 3-week treatment period (treatment period 1) during which Group A used Gum X and Group B used Gum S (2 gum pieces, 3 times daily after meals for 6 minutes). Both groups then underwent another 4-week washout period before entering treatment period 2 during which Group A used Gum S and Group B used Gum X for 3 weeks.

Sample collection: Saliva and plaque were collected from participants immediately before and after each treatment period (Figure 1). Subjects were instructed not to brush their teeth or use any other oral hygiene procedures at least 24 hours before sample collection, and not to eat or drink at least 1 hour before. For saliva collection, subjects chewed sterile paraffin wax and whole saliva produced was collected for 5 minutes in sterile tubes. The subject was asked to drool into the labelled 50ml collection tube (Falcon sterile, conical polypropylene tube with flat-top screw cap). This process was repeated multiple times in order to collect larger volumes of saliva (2-5 ml). The saliva was transferred via sterile pipettes into labelled sterile centrifuge tubes which were stored at -70˚C until use.

Supragingival plaque was collected with a curette from 2 molars (#16 and #36), 2 premolars (#24 and #44), and 2 incisors (#21 and #41); Plaque collection involved using a Gracey curette to remove all of the supragingival plaque from the buccal surface of the selected index tooth with as many strokes as necessary. The curette tip was immersed in the sterile DNase-free Tris-EDTA (TE) buffer in the centrifuge tube for 4-5 seconds. The face of the curette was wiped on the inside edge of the collection tube and then wiped off with sterile gauze so as to not let the buffer on the tip go into patient's mouth. The site was then immediately sampled again using the same procedure. The lid on the tube was replaced and then the tube shaken for 4-5 seconds in an attempt to maximize dispersion of the specimen in the fluid. The tube was immediately placed on ice in a Ziploc bag and stored at -70˚C until use. Samples were labelled by group (A/B), treatment period (1/2), gum used (X/S in the case of those samples collected at the end of a given treatment period) and type (saliva (s) or plaque (p)). Samples (n=232) were then shipped on dry ice to the J. Craig Venter Institute (JCVI) USA, La Jolla campus for DNA extraction and sequencing.

DNA extraction: Samples were thawed at 4˚C and vortexed thoroughly prior to DNA extraction from 500ul of saliva or plaque suspension using bead beating Lysing Matrix B tubes (MPBio Inc.), then lysozyme digest, phenol/chloroform isoamyl alcohol extraction and ethanol precipitation. Precipitated DNA was resuspended in 1x TE buffer.

Library Preparation and Sequencing: DNA from each sample was quantified using a Nanodrop spectrophotometer (Thermo Fisher Scientific, Inc, Waltham, MA). Amplicons were generated using adaptor and barcode ligated polymerase chain reaction (PCR) primers targeting the V4 region of the 16S rDNA gene (16S) and purified using Qiaquick PCR purification kits (Qiagen, Inc) following manufacturer's instructions. Purified amplicons were quantified using SybrGold (Thermo Fisher Scientific, Inc, Waltham, MA), normalized to ensure equimolar quantities of each sample, and pooled in preparation for Illumina MiSEQ sequencing. The 16S library pool was sequenced using the Illumina MiSEQ dual index 2x250bp V2 chemistry kit according to manufacturer's specifications.

16S RNA sequence data processing: Sequences for each sample were binned according to corresponding dual indices and exported as individual .fastq files using CASAVA v1.8.2 (Illumina Inc. La Jolla, CA). Sequences were processed to ensure that only quality sequences were retained, as stringent settings were kept to ensure no barcode mismatches were permitted during demultiplexing. Processed sequences were applied to the Infernal pipeline [35] for additional quality control (QC) checks. Bacterial sequences were taxonomically assigned based on the Genomic-based 16S ribosomal RNA Database (GRD; http://metasystems.riken.jp/grd/).

Statistical analyses. Distribution by age, sex and DMFT score for subjects in groups A and B were compared using independent-samples T- test, Pearson's Chi-Squared test and Wilcoxon rank sum test respectively, with a cut-off of p <0.05. To avoid possible sequence errors, operational taxonomic unit (OTU) count tables were filtered such that OTUs present in fewer than 0.1% in all samples were discarded. OTU tables were then transformed to relative abundances before community analyses were performed using the R statistical computing language (Cite R). Kruskal-Wallis test was used to assess statistical significance in microbial community composition across treatments. Wilcoxon test was used for pairwise comparison.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, subjects must have been 18 years and over, have had at least 20 teeth, provided written informed consent and been willing to comply with study procedures

Exclusion Criteria:

Subjects with systemic, infectious or inflammatory diseases or taking medicines, antibiotics or fluoride in the last month, habitual consumers of xylitol / sorbitol-containing products and mouth rinses, with abnormal salivary flow (<1ml / min), pregnant, on contraceptive pills, or with abnormal dietary habits were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2015-06-04 (Actual); Study Completion 2015-06-04 (Actual)

PRIMARY OUTCOMES:
Oral microbiome composition | 14 weeks
  Profile microbial communities of saliva and plaque based high-throughput sequencing of the 16S rRNA gene.

CONTACTS AND LOCATIONS:
Overall Officials: Reisha Rafeek, MSc, BDS, Principal Investigator — The University of The West Indies

IPD SHARING:
Plan to Share IPD: No